# **Evaluation of a Comprehensive School Health Programme in Zambia**

NCT number: (not yet assigned)

Unique Protocol ID: 264865

Dated: 7 December 2023

Participant information sheet and consent forms

#### **INFORMATION SHEET - HEADTEACHER**

Study Title: Evaluation of a school health program in Zambia

#### Who is carrying out this study and what is this study about?

This study is done by the University of Zambia (UNZA), the London School of Economics in the UK and the University of Virginia in the US.

The objective of the study is to measure the effects of a school health program run in some schools in six districts: Samfya, Mwense, Kawambwa, Masaiti, Chingola, Luanshya. We want to know if the program improves the health and learning of children. Your school has been chosen to take part in the study because it is either implementing some school health activities or it is currently in the comparison group but will introduce school health activities later.

# What does participation in this study involve?

If you agree to participate, we would need your support for two different activities involved in this study. *Activity 1:* School survey

We would like to ask you a few questions about your school, its infrastructure and staff. This will take approximately one hour 30 minutes to complete and will be organised at a time that is convenient for you. *Activity 2: Attendance spot check* 

We have a list of children whose attendance we would like to check at regular intervals. We would also like to choose two different classes (one Grade 6 and one Grade 7). For each one, we will copy the names of all children, then we will check who is at school today. We will also come back a few times this year (between 3 and 5 times) and we will repeat the same process in the same classes. For each class, this should not take more than 10 minutes.

#### Are there any disadvantages or benefits to me of taking part?

To compensate for your time and effort to take part in the study, you will receive Kw 50.

In addition, this study will provide useful information about the effects of the potential benefits of school health. Taking part in this study will not cause any harm to you.

#### Who will have access to the information I give?

- We will use the information you provide for this research project. All information collected about you will be kept private. We will keep all information about you safe and secure.
- Data may be sent to other study staff (in the UK, US) but this will be anonymised, meaning that your name
  and school name will be removed so that you cannot be recognised and your data will have a code
  number instead.
- We will share summaries of research findings with other researchers and government authorities through reports, presentations at meetings and publishing papers in scientific journals.
- At the end of the project, the data will be archived and made available to other researchers worldwide for research and to improve knowledge about health and education of school children. Your personal information will not be included and there is no way that you can be identified.

#### What will happen if I refuse to participate?

All participation in research is voluntary. You are free to decide if you want to take part or not. Even after agreeing, you can still change your mind at any time without any consequences, or choose to not answer specific questions if you are uncomfortable.

# What if I have any questions?

Do you have any questions? You are free to ask me any question about this research.

If you have any further questions about the study, you are free to contact the research team using the contacts below:

Professor Godfrey Biemba

National Health Research Authority (NHRA)

+260974770293

gbiemba@gmail.com

If you want to ask someone independent anything about this research please contact: ERES Converge

+26 095 515 5633

# **CONSENT FORM – HEADTEACHER**

# **Study Title:**

| Name of Researcher responsible for the project: Dr. Mylene Lagarde | | |
|---|---|---|
| Statement | Please initial each box | |
| I confirm that I have read and unders<br>above named study. I have had the of<br>questions and have these answered sa | | |
| I understand that my consent is voluit consent at any time without giving consequences. | | |
| I understand that the information I p repository or by sharing directly with identifiable from this information. | | |
| I agree to take part in the above named | | |
| Printed name of participant | Signature of participant | Date |

#### **INFORMATION SHEET - TEACHER**

Study Title: Evaluation of a school health program in Zambia

# Who is carrying out this study and what is this study about?

This study is done by the University of Zambia (UNZA), the London School of Economics in the UK and the University of Virginia in the US.

The objective of the study is to measure the effects of a school health program run in some schools in six districts: Samfya, Mwense, Kawambwa, Masaiti, Chingola, Luanshya. We want to know if the program improves the health and learning of children.

Your school has been chosen to take part in the study because it is either implementing some school health activities or it is currently in the comparison group but will introduce school health activities later.

# What does participation in this study involve?

If you agree to participate, we would like to ask you a few questions about your school, its infrastructure and staff. This will take approximately 45 minutes to complete and will be organised at a time that is convenient for you.

#### Are there any disadvantages or benefits to me of taking part?

To compensate for your time and effort to take part in the study, you will receive Kw 50.

In addition, this study will provide useful information about the effects of the potential benefits of school health. Taking part in this study will not cause any harm to you.

#### Who will have access to the information I give?

- We will use the information you provide for this research project. All information collected about you will be kept private. We will keep all information about you safe and secure.
- Data may be sent to other study staff (in the UK, US) but this will be anonymised, meaning that your name
  and school name will be removed so that you cannot be recognised and your data will have a code
  number instead.
- We will share summaries of research findings with other researchers and government authorities through reports, presentations at meetings and publishing papers in scientific journals.
- At the end of the project, the data will be archived and made available to other researchers worldwide for research and to improve knowledge about health and education of school children. Your personal information will not be included and there is no way that you can be identified.

#### What will happen if I refuse to participate?

All participation in research is voluntary. You are free to decide if you want to take part or not. Even after agreeing, you can still change your mind at any time without any consequences, or choose to not answer specific questions if you are uncomfortable.

#### What if I have any questions?

Do you have any questions? You are free to ask me any question about this research.

If you have any further questions about the study, you are free to contact the research team using the contacts below:

Professor Godfrey Biemba National Health Research Authority (NHRA) +260974770293 gbiemba@gmail.com

If you want to ask someone independent anything about this research please contact:

**ERES Converge** 

+26 095 515 5633

# **CONSENT FORM – TEACHER**

# **Study Title:**

Name of Researcher responsible for the project: Dr. Mylene Lagarde

| Statement | | Please initial each box |
|---|---|---|
| I confirm that I have read and under above named study. I have had the o questions and have these answered sa | | |
| I understand that my consent is volu consent at any time without giving consequences. | | |
| I understand that the information I prepository or by sharing directly with identifiable from this information. | | |
| I agree to take part in the above name | d study. | |
| Printed name of participant | Signature of participant | Date |
| Drivita di navo a finava a chitainina Ci | | |

#### **INFORMATION SHEET - PARENT (1)**

**Study Title:** Evaluation of a school health program in Zambia

#### Who is carrying out this study and what is this study about?

This study is done by the University of Zambia (UNZA), the London School of Economics in the UK and the University of Virginia in the US.

The objective of the study is to measure the effects of a school health program run in some schools in six districts: Samfya, Mwense, Kawambwa, Masaiti, Chingola, Luanshya. We want to know if the program improves the health and learning of children.

Your child has been chosen to take part in the study because s-he attends a school that is either introducing some school health activities now or is currently in the comparison group but will introduce them later.

#### What does participation in this study involve?

If you agree to participate, there are three different activities involved in this study. <u>Activity</u> <u>1: Interview with parent</u>

This interview will take approximately 30 minutes to complete and will be organised at a time that is convenient for you. We will ask a few questions about yourself and members of your household. This will be arranged in the next few days, probably at school. <u>Activity 2:</u> Interview with your child

This interview will take approximately 45 minutes to complete and will be organised at a time that is convenient for you. The interview will focus on your child's health and learning. We will also administer some tests to your child to monitor their learning throughout the program. This will be arranged in the next few days, probably at school. <u>Activity 3:</u> Symptom diaries

Next year, we will ask you to record over several weeks symptoms of diseases (e.g., fever, stomach pain) that your child may experience. We will also ask you to record if you seek care for any of this (either at home, in a pharmacy or somewhere else). We will provide a simple notebook to record all of this and arrange for collection at school.

#### Are there any disadvantages or benefits to me of taking part?

To compensate for your time and effort to take part in the study, you will receive Kw 50.

In addition, this study will provide useful information about the effects of the potential benefits of school health. Taking part in this study will not cause any harm to you or your child.

#### Who will have access to the information I give?

- We will use the information you provide for this research project. All information collected about you will be kept private. We will keep all information about you safe and secure.
- Data may be sent to other study staff (in the UK, US) but this will be anonymised, meaning that your name will be removed so that you cannot be recognised and your data will have a code number instead.
- We will share summaries of research findings with other researchers and government authorities through reports, presentations at meetings and publishing papers in scientific journals.
- At the end of the project, the data will be archived and made available to other researchers worldwide for research and to improve knowledge about health and education of school children. Your personal information will not be included and there is no way that you can be identified.

#### What will happen if I refuse to participate?

All participation in research is voluntary. You are free to decide if you want to take part or not. Even after agreeing, you can still change your mind at any time without any consequences, or choose to not answer specific questions if you are uncomfortable.

# What if I have any questions?

Do you have any questions? You are free to ask me any question about this research.

If you have any further questions about the study, you are free to contact the research team using the contacts below:

Professor Godfrey Biemba National Health Research Authority (NHRA) +260974770293 gbiemba@gmail.com

If you want to ask someone independent anything about this research please contact: ERES Converge +26 095 515 5633

| Learner name: | ID: | _ Gender: F / N | M Grade: 1 / 3 / 5 |
|---|---|---|---|
| CONSENT FORM – PARENT (1) | | | |
| Study Title: Evaluation of a school hea | . • | Languda | |
| Name of Researcher responsible for Statement | the project: Dr. Mylene | | Please initial each box |
| I confirm that I have read and understood the information sheet dated for the above named study. I have had the opportunity to consider the information, ask questions and have these answered satisfactorily. | | | . 15455 IIIIIII OUGII BOX |
| I understand that my consent is voluntary and that I am free to withdraw this consent at any time without giving any reason and without any negative consequences to me or my child. | | | |
| I understand that the information about me / my child provide may be shared via a public data repository or by sharing directly with other researchers, and that neither I nor my child or their school will not be identifiable from this information. | | | |
| I agree to me / my child taking part in the above named study. | | | |
| Printed name of participant | Signature of participant | | Date |
| Printed name of person obtaining Sig | gnature of person obtaini | ng consent Da | ate consent |

#### **INFORMATION SHEET - CHILD**

| _ | | _ | | |
|----|------|-----|-------|-----|
| I۳ | + | ٠A. | . Ati | ^ n |
| ш | LI C | λuι | ıcti | OH |

Good morning/afternoon. My name is [\_\_\_\_\_\_], and I am working for the "School Health Evaluation" study run by the University of Zambia (UNZA), the London School of Economics in the UK and the University of Virginia in the US.

#### Overview of the study

The objective of the study is to measure the effects of a school health program run in some schools.

#### What is involved?

If you agree to participate, we would like to ask you some questions about your health, your school, teachers, and your schoolwork. These questions should take about 30 minutes to complete.

# Confidentiality

The information I write down about you and other children will be kept safely locked up. When I tell other people or write an article about my research, I will not use your name so no one will know what you said. Remember there are no right or wrong answers.

#### **Voluntary participation**

Please talk this over with your parents before you decide whether to participate in the research study. We will also ask your parents or legal guardian if it is alright for you to take part in this study. But even if your parents say "yes" you can still decide not to do this.

You do not have to speak with me. It is okay if you decide you do not want to speak with me. Also, you can start to speak with me and then change your mind and stop at any time. No one will be mad at you. You can say no even if the headteacher said yes.

#### **Potential Benefits and Risks**

Nothing bad can happen if you decide to talk to us.

If you decide to participate in the study, you will help us learn more about what can be done to help students stay healthy in schools. We will also give you a little gift as a thank you.

#### **Questions**

You can ask any questions that you have about the study, and I will answer them for you.

If you have a question later, you can call me or contact at the following address:

Professor Godfrey Biemba National Health Research Authority (NHRA) +260974770293 gbiemba@gmail.com

# **ASSENT FORM - CHILD**

You and your parents will be given a copy of this form after you have signed it. Signing your name at the bottom means that:

- You have understood what I explained;
- You were able to ask questions if you wanted, and I answered them; You agree to be in this study.

| PARTICIPANT: | | |
|----------------|-----------|------|
| Name (Printed) | Signature | Date |
| RESEARCHER: | | |
| Name (Printed) | Signature | Date |

#### **INFORMATION SHEET - HEALTH FACILITY**

Study Title: Evaluation of a school health program in Zambia Who

#### is carrying out this study and what is this study about?

This study done by the University of Zambia (UNZA), the London School of Economics in the UK and the University of Virginia in the USA.

The objective of the study is to measure the effects of a school health program run in some schools in six districts: Samfya, Mwense, Kawambwa, Masaiti, Chingola, Luanshya. We want to know if the program improves the health and learning of children.

We are interested in finding out the perspectives of health workers and effects on the healthcare system.

Your facility has been chosen at random together with about 160 other facilities located in these six districts.

#### What does participation in this study involve?

If you agree to participate, we would like to interview you.

This interview will take approximately 45 minutes to complete and will be organised at a time that is convenient for you. The interview will focus on your experience, facility patient volume, waiting times, staff availability and expertise.

#### Are there any disadvantages or benefits to me of taking part?

This study will provide useful information about the effects of the potential benefits of school health. Taking part in this study will not cause any harm to you or affect your reputation or role within this health facility. We will never share the information you provide with your employer.

# Who will have access to the information I give?

- We will use the information you provide for this research project. All information collected about you will be kept private, safe and secure.
- With your permission, we will keep the data you give us until the end of the project (in 2026), after which we will remove personal information about you from our data servers. We may contact you again using these details before the end of 2026 and you can choose whether or not to speak to us again.
- Data will be sent to other study staff (in the UK, US) but this will be anonymised, meaning that your name and facility name will be removed so that you cannot be recognised and your data will have a code number instead.
- We will share the research results, as a summary across all 160 health facilities, with other researchers and government authorities in study reports, presentations and published papers in scientific journals.
- At the end of the project, the anonymised data will be archived and made available to other researchers worldwide for research and to improve knowledge about health and education. Your personal information will not be included and there is no way that you can be identified.

#### What will happen if I refuse to participate?

All participation in research is voluntary. You are free to decide if you want to take part or not. Even after agreeing, you can still change your mind at any time without any consequences, or choose to not answer specific questions if you are uncomfortable.

#### What if I have any questions?

Do you have any questions? You are free to ask me any question about this research.

If you have any further questions about the study, you are free to contact the research team using the contacts below:

Professor Godfrey Biemba National Health Research Authority (NHRA) +260974770293 gbiemba@gmail.com Professor Mylene Lagarde London School of Economics and Political Science +447595911011 m.lagarde@lse.ac.uk

If you want to ask someone independent anything about this research please contact: ERES Converge +26 095 515 5633

#### **CONSENT FORM - HEALTH FACILITY**

Study Title: Evaluation of a school health program in Zambia

| Name of Researcher responsible for the project: Professor Mylene Lagarde | | |
|---|---|---|
| Statement | | Please initial each box |
| I confirm that I have read and unders<br>above named study. I have had the op<br>questions and have these answered sa | | |
| I understand that my consent is volur consent at any time without giving consequences. | | |
| I understand that the information I prepository or by sharing directly with identifiable from this information. | | |
| I consent to my contact information be secure servers until 2026. I consent for to re-contact me. | | |
| I agree to take part in the above named | | |
| Drinted name of narticinant | Cionatura of narticinant | Data |
| Printed name of participant | Signature of participant | Date |

#### **INFORMATION SHEET - HEALTH WORKER**

Study Title: Evaluation of a school health program in Zambia

#### Who is carrying out this study and what is this study about?

This study done by the University of Zambia (UNZA), the London School of Economics in the UK and the University of Virginia in the USA.

The objective of the study is to measure the effects of a school health program run in some schools in six districts: Samfya, Mwense, Kawambwa, Masaiti, Chingola, Luanshya. We want to know if the program improves the health and learning of children.

We are interested in finding out the perspectives of health workers and effects on the healthcare system.

Your facility has been chosen at random together with about 160 other facilities located in these six districts.

#### What does participation in this study involve?

If you agree to participate, we would like to interview you.

This interview will take approximately 30 minutes to complete and will be organised at a time that is convenient for you. The interview will focus on your experience, your clinical knowledge and what you may know about the school health program.

#### Are there any disadvantages or benefits to me of taking part?

This study will provide useful information about the effects of the potential benefits of school health. Taking part in this study will not cause any harm to you or affect your reputation or role within this health facility. We will never share the information you provide with your employer.

# Who will have access to the information I give?

- We will use the information you provide for this research project. All information collected about you will be kept private, safe and secure.
- With your permission, we will keep the data you give us until the end of the project (in 2026), after which we will remove personal information about you from our data servers. We may contact you again using these details before the end of 2026 and you can choose whether or not to speak to us again.
- Data will be sent to other study staff (in the UK, US) but this will be anonymised, meaning that your name and facility name will be removed so that you cannot be recognised and your data will have a code number instead.
- We will share the research results, as a summary across all 160 health facilities, with other researchers and government authorities in study reports, presentations and published papers in scientific journals.
- At the end of the project, the anonymised data will be archived and made available to other researchers worldwide for research and to improve knowledge about health and education. Your personal information will not be included and there is no way that you can be identified.

#### What will happen if I refuse to participate?

All participation in research is voluntary. You are free to decide if you want to take part or not. Even after agreeing, you can still change your mind at any time without any consequences, or choose to not answer specific questions if you are uncomfortable.

#### What if I have any questions?

Do you have any questions? You are free to ask me any question about this research.

If you have any further questions about the study, you are free to contact the research team using the contacts below:

Professor Godfrey Biemba National Health Research Authority (NHRA) +260974770293 gbiemba@gmail.com Professor Mylene Lagarde London School of Economics and Political Science +447595911011 m.lagarde@lse.ac.uk

If you want to ask someone independent anything about this research please contact: ERES Converge +26 095 515 5633

#### **CONSENT FORM – HEALTH WORKER**

Study Title: Evaluation of a school health program in Zambia

| Name of Researcher responsible for the project: Professor Mylene Lagarde | | |
|---|---|---|
| Statement | | Please initial each box |
| I confirm that I have read and unders<br>above named study. I have had the op<br>questions and have these answered sa | | |
| I understand that my consent is volur consent at any time without giving consequences. | | |
| I understand that the information I prepository or by sharing directly with identifiable from this information. | | |
| I consent to my contact information be secure servers until 2026. I consent for to re-contact me. | | |
| I agree to take part in the above named | | |
| Drinted name of narticinant | Cionatura of narticinant | Data |
| Printed name of participant | Signature of participant | Date |